CLINICAL TRIAL: NCT02732158
Title: Feasibility of Novel Laboratory Methods for Use in Nutrition Studies
Brief Title: Novel Laboratory Methods in Nutrition Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL27
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Novel laboratory methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition Products (Experimental): Two servings per day of the sachet study product mixed with water; 1 carotenoid capsule per day
  Interventions: Other: Nutrition Products

INTERVENTIONS:
Other: Nutrition Products — a sachet containing AN777and amino acids; a carotenoid capsule

SUMMARY:
This prospective, nonrandomized, feasibility study will compare laboratory measures at the beginning and end of the study period in adults consuming a nutritional study product.

ELIGIBILITY:
Inclusion Criteria:

* Participant must agree to refrain from taking supplements other than study product.
* Participant states willingness to follow protocol as described, including consumption of study product per protocol, performing finger stick/DBS on Day 60 and completing any forms needed throughout the study.

Exclusion Criteria:

* Body Mass Index (BMI) > or equal to 35 kg/m2
* Has planned elective surgery requiring 2 or more days of hospitalization during the entire study
* Has stated active malignant disease
* Has a known history of chronic renal parenchymal disease
* Has a known history of severe liver disease/liver failure
* Has any psychiatric disorders that would interfere with study product consumption or compliance with the study procedures
* Known allergy or intolerance to any study product ingredient
* Participation in another study that has not been approved as a concomitant study

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Comparison of lab values from venipuncture and DBS methods | Baseline
  Correlation and difference in baseline levels of AN777 and carotenoids between samples collected through venipuncture and fingerstick on dried blood spot (DBS) cards.

SECONDARY OUTCOMES:
Change in AN777 | Baseline to Day 60
Change in carotenoids | Baseline to Day 60
Compliance of study product consumption | Baseline to Day 60
  Subject Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Alish, PhD, RD, Study Chair — Abbott Nutrition
Locations (1):
- Texas A&M University, Center for Translation Research in Aging and Longevity, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No